CLINICAL TRIAL: NCT02934503
Title: A Phase II Study of Pembrolizumab and Dynamic PD-L1 Expression in Extensive Stage Small Cell Lung Cancer (SCLC)
Brief Title: Study of Pembrolizumab and Chemotherapy With or Without Radiation in Small Cell Lung Cancer (SCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated as the standard of care for small cell lung cancer changed in 2018 to include immunotherapy in the front line setting, making this study no longer clinically relevant.
Sponsor: NYU Langone Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01031
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Chemotherapy; PD-L1; Thoracic radiotherapy; PD-1; MK-3475
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pembrolizumab; Cisplatin; Carboplatin; Etoposide; etoposide phosphate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cisplatin or carboplatin, Etoposide, Pembrolizumab & Radiation (Experimental): Cohort A: cisplatin (75 mg/m^2) + carboplatin (AUC 6) + etoposide (100mg/m^2) for four to six, 3-week cycles + pembrolizumab (200 mg) followed by radiation. Pembrolizumab will be started with first cycle of chemotherapy and continued for up to 2 years.
  Cohort B: Pembrolizumab (200 mg) will be added to standard therapy with cisplatin (75 mg/m2) or carboplatin (AUC 6) and etoposide (100 mg/m2) (and radiation, if appropriate), after one 3- week cycle of standard therapy and continued for up to 2 years.
  Cohort C: 200 mg IV infusion of Pembrolizumab every 3 weeks over about 30 minutes after completion of standard chemotherapy with cisplatin (75 mg/ m2) and etoposide (100 mg/m2). Treatment with pembrolizumab will continue for up to 2 years.
  Cohort D: Pembrolizumab 200 mg IV infusion every 3 weeks in vein after completion of standard chemotherapy and radiation. Pembrolizumab will start within 6 weeks of completing radiation therapy and continue for up to 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg IV fixed dose every 3 weeks until progression or for up to 2 years of therapy.
  Other Names: Keytruda
Drug: Cisplatin — 75 mg/m2
  Other Names: Platinol
Drug: Carboplatin — AUC 6
  Other Names: Paraplatin
Drug: Etoposide — IV every 3 weeks for up to 6 cycles (minimum of 4 cycles, maximum of 6).
  Other Names: Etopophos
Radiation: Radiation therapy — Thoracic radiotherapy will be given per institutional standards(dose and duration may vary for individual participants).

SUMMARY:
This trial is to assess the efficacy of pembrolizumab added to concurrent chemotherapy with or without radiation therapy in patients with small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
SCLC provides an opportune setting to evaluate the potential importance of variability in PD-L1 expression and its influence on optimizing timing and efficacy of checkpoint inhibition. All extensive stage SCLC patients are treated with chemotherapy and recent data suggests added benefit to consolidation thoracic radiation. A prior study of patients with known PD-L1 expression showed a 35% response rate. That study used archival specimens and found a 29% PD-L1 positivity rate (at 1% level) suggesting that the expression level and prevalence could be higher (and response rate/outcome therefore potentially better) in patients who have previously had chemotherapy or radiation. The proposed study seeks to evaluate pembrolizumab therapy initiated at different times during the course of SCLC treatment: a) up front, in conjunction with initiation of chemotherapy, b) starting after one cycle of chemotherapy, c) starting after completion of 1st line chemotherapy (4-6 cycles), d) starting after completion of consolidation thoracic radiation therapy and/or prophylactic cranial irradiation (PCI). Treatment with pembrolizumab will be preceded by biopsy for evaluation of PD-L1 expression with correlative evaluation of changes in PD-L1 expression (relative to diagnostic biopsy) and changes in other tissue- and blood-based biomarkers and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed small cell lung carcinoma not amenable to initial concurrent radiotherapy (extensive-stage disease).
* Participants may have evaluable or measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Participants in cohort B must have completed 1 cycle of systemic chemotherapy. Therapy with the combination must start no sooner than 3 weeks from the last dose of chemotherapy and no later than 5 weeks from the last dose of chemotherapy. Participants in cohort B must not have had progression of disease prior to the start of therapy.
* Participants in cohort C must have completed systemic therapy (4-6 cycles cisplatin or carboplatin + etoposides) and NOT be a candidate for consolidation thoracic radiotherapy or PCI. Participants in cohort C must initiate therapy with pembrolizumab within 6 weeks of the last dose of chemotherapy (therapy must not start within 2 weeks from the last dose). Participants in cohort C must not have had progression of disease prior to the start of therapy.
* Participants in cohort D must have completed systemic therapy AND have completed either consolidation thoracic radiotherapy or PCI or both completed either consolidation thoracic radiotherapy or PCI or both. Participants in cohort D must initiate therapy with pembrolizumab within 6 weeks of the last dose of radiation. Therapy must not start within 2 weeks from the last dose. Consolidation radiotherapy dose must NOT be more than 3000 centigray (cGy). Participants in cohort D must not have had progression of disease prior to the start of therapy.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%)
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function during screening and on Cycle 1, day 1 as defined below.

  * Adequate Organ Function Laboratory Values
* System Laboratory Value Hematological
* Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL)
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)

Renal

* Serum creatinine OR Measured or ≤1.5 X upper limit of normal (ULN) OR calculated creatinine ≥60 mL/min for subject with creatinine clearance (GFR can also be used levels >1.5X institutional ULN in place of creatinine or CrCl)

Hepatic

* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and Alanine transaminase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin >2.5 mg/dL

Coagulation

* International Normalized Ratio ≤1.5 X ULN unless subject is receiving (INR) or Prothrombin Time (PT) anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin ≤1.5 X ULN unless subject is receiving Time (aPTT) anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Availability of a diagnostic or pre-chemotherapy tissue biopsy is required (cytologic specimens or bone biopsies not accepted). This biopsy must be within 6 weeks of starting initial therapy. A minimum of 205 μm slides or block is required.
* Participants in cohorts B-D must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen within 4 weeks to initiation of treatment and AFTER the last dose of any prior therapy.
* Participants with treated brain metastases are allowed. Radiation must be completed at least 2 weeks prior to pembrolizumab dosing and participants must not require ongoing steroids. Participants with untreated brain metastases that are all <5 mm with no clinical symptoms or vasogenic edema may be allowed on study on a case-by-case basis on discussion with sponsor. These participants will require MRI monitoring every 6 weeks to ensure stability.
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason and because the chemotherapy and radiation also used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) or be surgically sterile prior to study entry and for the duration of study participation. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of chemotherapy, radiation, and pembrolizumab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants in cohort A may not have had prior therapy for their disease. Participants in cohort B may not have had more than 1 cycle of systemic therapy (cisplatin or carboplatin + etoposide). Participants in cohort C and D should not have had more than one prior regimen of chemotherapy.
* For participants entering cohorts C or D, prior treatment-related toxicities should have resolved to grade 1 or baseline (with the exception of anemia (as per inclusion criteria, alopecia, and neuropathy (< grade 2 allowed).
* Participants who have had a CR after pre-study therapy are not eligible for study.
* No thoracic radiation > 3000 cGy allowed.
* Prior radiation or surgery must have completed at least 2 weeks prior to initiation of therapy and all toxicities or complications from these must have resolved to baseline or grade 1 prior to starting therapy (with the exception of anemia (as per inclusion criteria, alopecia, and neuropathy (< grade 2 allowed).
* No stroke, myocardial infarction, or major surgery within 3 months of starting on therapy
* Participants who are receiving any other investigational agents or have received investigational therapy or any anti-cancer monoclonal antibody (mAB) within 4 weeks prior to the 1st dose of pembrolizumab.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of non-infectious pneumonitis which required steroids, or any evidence of current, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, cisplatin, carboplatin, or etoposide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C Virus (HCV) (e.g., HCV RNA [qualitative] is detected).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has received a live vaccine within 30 days of planned start of study therapy Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist are live attenuated vaccines, and are not allowed.
* Has a known additional malignancy that is progressing or requires active treatment or has required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or in situ bladder cancer.
* Has a paraneoplastic syndrome other than SIADH (hyponatremia).
* Evidence of interstitial lung disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Sabari, MD,, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated as the standard of care for small cell lung cancer changed in 2018 to include immunotherapy in the front line setting, making this study no longer clinically relevant. Due to this change in standard of care practice, the study was closed. It only accrued 5 participants - randomization/proper crossover assignment was not performed; therefore, data is not presented "per arm".
Groups:
- Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation: Cohort A: cisplatin (75 mg/m^2) + carboplatin (AUC 6) + etoposide (100mg/m^2) for four to six, 3-week cycles + pembrolizumab (200 mg) followed by radiation. Pembrolizumab will be started with first cycle of chemotherapy and continued for up to 2 years.
  Cohort B: Pembrolizumab (200 mg) will be added to standard therapy with cisplatin (75 mg/m2) or carboplatin (AUC 6) and etoposide (100 mg/m2) (and radiation, if appropriate), after one 3- week cycle of standard therapy and continued for up to 2 years.
  Cohort C: 200 mg IV infusion of Pembrolizumab every 3 weeks over about 30 minutes after completion of standard chemotherapy with cisplatin (75 mg/ m2) and etoposide (100 mg/m2). Treatment with pembrolizumab will continue for up to 2 years.
  Cohort D: Pembrolizumab 200 mg IV infusion every 3 weeks in vein after completion of standard chemotherapy and radiation. Pembrolizumab will start within 6 weeks of completing radiation therapy and continue for up to 2 years.
  Pembrolizumab: 200 mg IV fixed dose every 3 weeks until progression or for up to 2 years of therapy.
  Cisplatin: 75 mg/m2
  Carboplatin: AUC 6
  Etoposide: IV every 3 weeks for up to 6 cycles (minimum of 4 cycles, maximum of 6).
  Radiation therapy: Thoracic radiotherapy will be given per institutional standards(dose and duration may vary for individual participants).
Period: Overall Study
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Started | 5
Completed | 1
Not Completed | 4
Not completed — progression of disease | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This study was terminated as the standard of care for small cell lung cancer changed in 2018 to include immunotherapy in the front line setting, making this study no longer clinically relevant. Due to this change in standard of care practice, the study was closed. It only accrued 5 participants - randomization/proper crossover assignment was not performed; therefore, data is not presented "per arm".
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 68 [59 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in PD-L1 Expression Status as Determined by Immunohistochemistry in Pretreatment and Archival Samples
Time Frame: up to 5 months
Population: This study was terminated as the standard of care for small cell lung cancer changed in 2018 to include immunotherapy in the front line setting, making this study no longer clinically relevant. Due to this change in standard of care practice, the study was closed. It accrued 5 patients and therefore there is insufficient data to report on any of the outcomes/endpoints.
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Progression-free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause
Time Frame: up to 6 months
Population: as for outcome 1
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: up to 9 months
Population: as for outcome 1
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Evaluation Using Response Evaluation Criteria In Solid Tumors (RECIST)
Time Frame: at 6 weeks
Population: as for outcome 1
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Evaluation Using Response Evaluation Criteria In Solid Tumors (RECIST)
Time Frame: at 12 weeks
Population: as for outcome 1
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 months
Description: This study was terminated as the standard of care for small cell lung cancer changed in 2018 to include immunotherapy in the front line setting, making this study no longer clinically relevant. Due to this change in standard of care practice, the study was closed. It only accrued 5 participants - randomization/proper crossover assignment was not performed; therefore, data is not presented "per arm".
Arm/Group | Cisplatin or Carboplatin, Etoposide, Pembrolizumab & Radiation
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02934503/Prot_SAP_000.pdf